CLINICAL TRIAL: NCT05456191
Title: A Phase IIIb, Multi-center, Open-label, Randomized Study of Tolerability and Efficacy of Oral Asciminib Versus Nilotinib in Patients With Newly Diagnosed Philadelphia Chromosome Positive Chronic Myelogenous Leukemia in Chronic Phase.
Brief Title: A Study to Investigate Tolerability and Efficacy of Asciminib (Oral) Versus Nilotinib (Oral) in Adult Participants (≥18 Years of Age) With Newly Diagnosed Philadelphia Chromosome Positive Chronic Myelogenous Leukemia in Chronic Phase (Ph+ CML-CP)
Acronym: ASC4START
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABL001J12302; 2024-510947-71-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT04360005 (Available)
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Philadelphia Chromosome-Positive Chronic Myeloid Leukemia
Keywords: Asciminib (ABL001); Abelson proto-oncogene (ABL); newly diagnosed Chronic Myelogenous Leukemia (CML); Chronic Myeloid Leukemia (CML); Chronic Myelocytic Leukemia (CML); Chronic Granulocytic Leukemia (CGL); cancer of the white blood cells; clonal bone marrow stem cell disorder proliferation of mature granulocytes; Chronic Myeloproliferative Disorders; Philadelphia chromosome; Nilotinib; Leukemia; Phase 3; Tyrosine Kinase Inhibitor (TKI); Treatment Free Remission (TFR); Treatment Re-initiation (TRI)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders; Philadelphia Chromosome; Leukemia | interventions — asciminib; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Asciminib (Experimental): Participants received asciminib 80 mg once a day (QD).
  Interventions: Drug: Asciminib
- Nilotinib (Active Comparator): Participants will receive nilotinib 300 mg BID
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Asciminib — Asciminib 80 mg QD administered under fasting conditions.
  Other Names: ABL001
  Arms: Asciminib
Drug: Nilotinib — Nilotinib 300 mg twice a day (BID) was administered under fasting conditions.
  Arms: Nilotinib

SUMMARY:
The primary purpose of this study was to assess the tolerability of oral asciminib (80 mg QD) in comparison with that of the second generation (2G) Tyrosine Kinase Inhibitor (TKI) nilotinib (300 mg BID), in adult patients with newly diagnosed Positive Chronic Myelogenous Leukemia in Chronic Phase (Ph+ CML-CP).

DETAILED DESCRIPTION:
Participants were randomized in the study in a 1:1 ratio to asciminib or nilotinib. No crossover of study treatment across arms were allowed.

Randomization was stratified based on European Treatment Outcome Study (EUTOS) long-term survival (ELTS) score (low versus intermediate versus high) to help achieve a balance between the treatment arms.

The primary analysis was performed when approximately 65 discontinuations of either study treatment due to Adverse Event (AE) occured.

Eligible participants on both arms could choose to participate in an optional 2-year Treatment Free Remission (TFR) Phase. Participants with loss of Major Molecular Response (MMR) during TFR Phase were to enter the Treatment Re-initiation (TRI) Phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male or female patients ≥ 18 years of age.
* Patients with CML-CP within 3 months of diagnosis.
* Diagnosis of CML-CP (European Leukemia Network [ELN] 2020 criteria) with cytogenetic confirmation of the Philadelphia (Ph) chromosome. A cryptic Ph chromosome should be confirmed by metaphase Fluorescence in situ Hybridization (FISH)

  * Documented chronic phase CML will meet all the below criteria (Baccarani et al 2013):
  * < 15% blasts in peripheral blood and bone marrow,
  * < 30% blasts plus promyelocytes in peripheral blood and bone marrow,
  * < 20% basophils in the peripheral blood,
  * Platelet (PLT) count ≥ 100 x 109/L (≥ 100,000/mm3),
  * No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly.
* Evidence of typical BCR::ABL1 transcript [e14a2 and/or e13a2] which is amenable to standardized RQ-PCR quantification by the central laboratory assessment. However, if a local qualitative assay, validated according to local regulation, from an accredited local laboratory has confirmed evidence of typical BCR::ABL1 transcript [e14a2 and/or e13a2], these results can be used for eligibility if the central Real Time Quantitative Polymerase Chain Reaction (RQ-PCR) results arrived are not available at the time of randomization.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate end organ function as defined by:

  • Total bilirubin (TBL) < 3 x Upper Limit of Normal (ULN); patients with Gilbert's syndrome may only be included if TBL ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN,
  * Creatinine Clearance (CrCl) ≥ 30 milliliters per minute (mL/min) as calculated using Cockcroft-Gault formula, Serum lipase ≤ 1.5 x ULN. For serum lipase > ULN - ≤ 1.5 x ULN, value must be considered not clinically significant and not associated with risk factors for acute pancreatitis.
* Patients must have the following laboratory values within normal limits or corrected to within normal limits with supplements prior to randomization:

  * Potassium (potassium increase of up to 6.0 mmol/L is acceptable if associated with CrCl* ≥ 90 mL/min)**,
  * Total calcium (corrected for serum albumin); (calcium increase of up to 12.5 mg/dl or 3.1 mmol/L is acceptable if associated with CrCl* ≥ 90 mL/min),
  * Magnesium (magnesium increase of up to 3.0 mg/dL or 1.23 mmol/L if associated with CrCl* ≥ 90 mL/min),
  * For patients with mild to moderate renal impairment (CrCl* ≥ 30 mL/min and <90 mL/min) - potassium, total calcium (corrected for serum albumin) and magnesium should be within normal limits or corrected to within normal limits with supplements prior to randomization.

    * CrCl as calculated using Cockcroft-Gault formula.

      * pseudohyperkaliemia in case of thrombocytosis is not an exclusion criterion.

Inclusion Criteria for optional Treatment Free Remission (TFR) Phase:

* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
* A minimum of 3 years (156 weeks) of treatment on study, up-to maximum of 5 years (260 weeks) of treatment.
* Sustained MR4.5 (BCR:ABL1 ≤0.0032% IS) for at least 1 year (≥52 weeks) immediately prior to entry into the TFR Phase, defined as 5 consecutive (every 12 weeks) central laboratory RQ-PCR assessments at MR4.5 or below for the course of at least a year. Entry into TFR Phase should be at an unscheduled visit or next scheduled visit no later than 12 Weeks from the last RQ-PCR assessment date at MR4.5 or lower.
* Separate signed informed consent must be obtained prior to participation in the TFR Phase.

Key Exclusion Criteria:

* Previous treatment of CML with any other anticancer agents including chemotherapy and/or biologic agents or prior stem cell transplant, with the exception of hydroxyurea and/or anagrelide.
* Known cytopathologically confirmed central nervous system (CNS) infiltration (in absence of suspicion of CNS involvement, lumbar puncture not required).
* Impaired cardiac function or cardiac repolarization abnormality including but not limited to any one of the following:

  • History of myocardial infarction (MI), angina pectoris, coronary artery bypass graft (CABG) within 6 months prior to starting study treatment.

  • Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II and third degree AV block).
  * QT interval corrected by Fridericia's formula (QTcF) ≥ 450 ms on the average of three serial baseline ECG (using the QTcF formula). If QTcF ≥ 450 ms and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTcF.
  * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

    * Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
    * Concomitant medication(s) with a "Known risk of Torsades de Pointes" per crediblemeds.org that cannot be discontinued or replaced 7 days prior to starting study treatment by safe alternative medication.
    * Inability to determine the QTcF interval.
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the Investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes, active or uncontrolled infection; uncontrolled arterial or pulmonary hypertension, uncontrolled clinically significant hyperlipidemia).
* History of significant congenital or acquired bleeding disorder unrelated to cancer.
* Major surgery within 4 weeks prior to study entry or patients who have not recovered from prior surgery.
* History of other active malignancy within 3 years prior to study entry with the exception of previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively.
* History of acute pancreatitis within 1 year prior to randomization or medical history of chronic pancreatitis.
* History of chronic liver disease leading to severe hepatic impairment, or ongoing acute liver disease.
* Known history of chronic Hepatitis B (HBV), or chronic Hepatitis C (HCV) infection. Testing for Hepatitis B surface antigen (HBs Ag) and Hepatitis B core antibody (HBc Ab/anti HBc) will be performed at screening. If anti-HBc is positive, HBV-DNA (deoxyribonucleic acid) evaluation will be carried out at screening. A patient having positive HBV-DNA will not be enrolled in the study. Also, a patient with positive HBsAg will not be enrolled in the study. HCV Ab testing will also be performed at screening. For details on the criteria see Appendix 10.4
* History of Human Immunodeficiency Virus (HIV) unless well-controlled on a stable dose of anti-retroviral therapy at the time of screening.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study treatment (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery).
* Participation in a prior investigational study within 30 days prior to randomization or within 5 half-lives of the investigational product, whichever is longer.
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for a period of time after stopping study medication. For asciminib, this period of time is 3 days after last dose; if local regulations or locally approved prescribing information differ from the protocol required duration of contraception, the longer duration must be followed and the same requirements will be described in the Informed Consent Form (ICF). Participants taking nilotinib should be willing to follow contraception requirements in the locally-applicable prescribing information for nilotinib.

Highly effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or total hysterectomy or bilateral salpingectomy, at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Male partner's sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participant
* Use of oral, (estrogen and progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.

In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Women are considered post-menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate history of vasomotor symptoms). Women are considered not of child bearing potential if they are post-menopausal or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral salpingectomy at least six weeks prior to enrollment on the study. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered to be not of child bearing potential.

Sexually active males taking study treatment do not require contraception. 16. Known hypersensitivity to the study treatment. Note: The Investigator has the discretion to include/exclude a patient in the study, who will be found to have symptoms representative of coronavirus disease of 2019 (COVID-19) or tested positive for COVID-19 during the screening phase. Such patients should be managed as per the country specific guidelines related to COVID-19. For patients who test positive for COVID-19, re-testing is recommended before initiating study treatment.

Exclusion Criteria for optional Treatment Free Remission (TFR) Phase:

• Participants in the TRI Phase cannot re-enter the TFR Phase for second attempt TFR.

Exclusion criteria for Treatment Re-initiation (TRI) Phase

• In case of a pregnancy during the TFR Phase, the pregnant woman must be discontinued from the study upon loss of MMR (>0.1% BCR::ABL1 IS at a single assessment) and cannot enter the TRI phase.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2031-07-07 (Estimated)

PRIMARY OUTCOMES:
Time to discontinuation of study treatment due to adverse event (TTDAE). | From date of first dose to date of treatment discontinuation due to AE, assessed up to 5 years
  TTDAE is defined as the time from the date of first dose of study treatment to the date of discontinuation of study treatment due to adverse event (AE).

SECONDARY OUTCOMES:
Percentage of participants with Major Molecular response (MMR) at scheduled data collection time points | approximately 7.5 years
  MMR will be assessed using fusion gene of the BCR and ABL genes (BCR-ABL) transcript levels measured by realtime quantitative polymerase chain reaction.
  The percentage of participants with MMR at each time point will be assessed.
Percentage of participants with Major Molecular response (MMR) by scheduled data collection time points | approximately 7.5 years
  MMR will be assessed using BCR-ABL transcript levels measured by realtime quantitative polymerase chain reaction.
  The percentage of participants who meet the criteria for having achieved the endpoint (MMR) at or before the specified visit will be calculated.
Percentage of participants with MR4.0 at scheduled data collection time points | approximately 7.5 years
  MR4.0 will be assessed using BCR-ABL transcript levels measured by realtime quantitative polymerase chain reaction.
  The percentage of participants with MR4.0 at each time point will be assessed.
Percentage of participants with MR4.0 by scheduled data collection time points | approximately 7.5 years
  MR4.0 will be assessed using BCR-ABL transcript levels measured by realtime quantitative polymerase chain reaction.
  The percentage of participants who meet the criteria for having achieved the endpoint (MR4.0) at or before the specified visit will be calculated
Percentage of participants with MR4.5 at scheduled data collection time points | approximately 7.5 years
  MR4.5 will be assessed using BCR-ABL transcript levels measured by realtime quantitative polymerase chain reaction.
  The percentage of participants with MR4.5 at each time point will be assessed.
Percentage of participants with MR4.5 by scheduled data collection time points | approximately 7.5 years
  MR4.5 will be assessed using BCR-ABL transcript levels measured by realtime quantitative polymerase chain reaction.
  The percentage of participants who meet the criteria for having achieved the endpoint (MR4.5) at or before the specified visit will be calculated
Percentage of participants with Complete Hematological response (CHR) at scheduled data collection time points | approximately 7.5 years
  Hematologic response will be assessed by complete blood count and physical examination at each visit.
  The percentage of participants with CHR at each time point will be assessed.
Percentage of participants with Complete Hematological response (CHR) by scheduled data collection time points | approximately 7.5 years
  Hematologic response will be assessed by complete blood count and physical examination at each visit.
  The percentage of participants who meet the criteria for having achieved the endpoint (CHR) at or before the specified visit will be calculated
Percentage of participants with BCR::ABL1 ratio ≤1% at scheduled data collection time points | approximately 7.5 years
  The percentage of participants who meet the criteria for having achieved BCR::ABL1 ratio ≤1% at the specified visit will be calculated
Percentage of participants with BCR::ABL1 ratio ≤1% by scheduled data collection timepoints | approximately 7.5 years
  The percentage of participants who meet the criteria for having achieved BCR::ABL1 ratio ≤1% at or before the specified visit will be calculated
Duration of MMR | approximately 7.5 years
  Duration of MMR is defined as the time between the date of the first documented achievement MMR and the earliest date of loss of MMR, treatment failure, progression to AP/BC, or CML-related death.
Duration of MR4.0 | approximately 7.5 years
  Duration of MR4.0 is defined as the time between the date of the first documented achievement MR4 and the earliest date of loss of MR4, treatment failure, progression to AP/BC, or CML-related death
Duration of MR4.5 | approximately 7.5 years
  Duration of MR4.5 is defined as the time between the date of the first documented achievement MR4.5 and the earliest date of loss of MR4.5, treatment failure, progression to AP/BC, or CML-related death.
Time to first MMR | approximately 7.5 years
  Time to first MMR is defined as the time from the date of randomization to the date of the first documented occurrence of MMR.
Time to first MR4.0 | approximately 7.5 years
  Time to first MR4.0 is defined as the time from the date of randomization to the date of the first documented occurrence of MR4.
Time to first MR4.5 | approximately 7.5 years
  Time to first MR4.5 is defined as the time from the date of randomization to the date of the first documented occurrence of MR4.5.
Time to treatment failure (TTF). | approximately 7.5 years
  TTF is defined as the time from date of randomization to the first/earliest documented date of any of the following events:
  * Treatment failure per European leukemia network (ELN) criteria,
  * Confirmed loss of MMR (in 2 consecutive tests) at any time while on study treatment,
  * Discontinuation from study treatment due to any reason
Event free survival (EFS) | approximately 7.5 years
  EFS is defined as the time from the date of the first dose of study treatment to the earliest occurrence of treatment failure, confirmed lost of MMR, discontinuation due to AE, progression to AP/BC, and death from any cause.
Progression free survival (PFS). | approximately 7.5 years
  PFS is defined as the time from the date of randomization to the earliest occurrence of progression to AP/BC or death from any cause.
Overall survival (OS). | approximately 7.5 years
  OS is defined as the time from the date of randomization to the date of death from any cause.
Time to treatment discontinuation (TTD) due to selected reasons | approximately 7.5 years
  TTD is the time from the date of first dose of study treatment to the date of discontinuation of study treatment due to lack of efficacy, treatment failure, disease progression, suboptimal response or death
Change from baseline in overall scores and individual scales of the European organization for research and treatment of cancer - quality of life questionnaire (EORTC QLQ-C30) | approximately 7.5 years
  Change from baseline in Overall Scores and individual domains of the EORTC QLQ-C30. The EORTC QLQ-C30 contains 30 items and is composed of both multi-item scales and single-item measures based on the participant's experience over the past week. These include five functional scales (physical, role, emotional, cognitive and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/QoL scale.
Change from baseline in overall scores and individual scales of the European organization for research and treatment of cancer CML module (EORTC QLQ-CML24) | approximately 7.5 years
  Change from baseline in Overall Scores and individual domains of the EORTC QLQ-CML24. The EORTC QLQ-CML24 assesses specific concepts relevant to the experience of patients with CML. The QLQ-CML24 has 24 items which assess symptom burden, impact on daily life and on worry/mood, body image problems, and satisfaction with care and with social life based on the participant's experience over the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (110):
- United States (9):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Illinois Cancer Care, Peoria, Illinois
  - Regions Hospital, Saint Paul, Minnesota
  - Messino Cancer Centers, Asheville, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Williamette Cancer Center, Eugene, Oregon
  - Texas Oncology P A, Bedford, Texas
  - Texas Oncology PA Bedford, Bedford, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, CABA
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (2):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Plzen Bory
  - Novartis Investigative Site, Prague
- France (13):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (31):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Paderborn, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
- Greece (4):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Eger
- India (5):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
  - Novartis Investigative Site, Rishikesh, Uttarakhand
- Italy (5):
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Novartis Investigative Site, Amman, Jordan
- Malaysia (4):
  - Novartis Investigative Site, Alor Star, Kedah
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Petaling Jaya, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Novartis Investigative Site, Dordrecht, South Holland, Netherlands
- Novartis Investigative Site, Khoudh, Oman
- Romania (6):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Târgu Mureş, Mureș County
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Sibiu
  - Novartis Investigative Site, Timișoara
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Bratislava, Slovakia
- South Africa (2):
  - Novartis Investigative Site, Johannesburg, Gauteng
  - Novartis Investigative Site, Pretoria, Gauteng
- South Korea (2):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggi-do
- Novartis Investigative Site, Geneva, Switzerland
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, Abu Dhabi, United Arab Emirates
- United Kingdom (4):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Gloucester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newport

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com